CLINICAL TRIAL: NCT06366178
Title: Evaluation of the Safety and Effectiveness of a Medical Device Aimed at Guiding Orbito-naso-frontal Band Surgery, for the Treatment of Craniostenoses
Brief Title: EPBONF : Evaluation of the Safety and Effectiveness of a Medical Device Aimed at Guiding Orbito-naso-frontal Band Surgery, for the Treatment of Craniostenoses
Acronym: EPBONF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/864
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Craniosynostoses
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- reshaping the orbito-naso-frontal band with a guide (Experimental)
  Interventions: Device: BONFIX system

INTERVENTIONS:
Device: BONFIX system — The device corresponds to a customized, single-use surgical guide (Class IIa medical device), with a set of different sizes, adapted to the fronto-zygomatic distance (FDZ) measurement, in order to enable better conformation of the orbito-naso-frontal bandeau during surgery for anterior craniostenosis, an ideal conformation that could lead to optimal symmetry and adapted to the morphology of the upper third of infants.
  The surgeon conforms the orbito-naso-frontal bandeau by adapting the advancement between the device supports according to the FDZ and then positioning it directly on the surgical guide.

SUMMARY:
Craniostenosis is a congenital disorder caused by early fusion of the cranial sutures between the skull bones, resulting in orbito-naso-frontal deformities. The damage is primarily aesthetic, but intracranial hypertension may also be observed.

The treatment of craniostenosis involves surgery, to restore harmonious growth between the skull bones and the brain, and proper development of the latter.

There are various surgical techniques for correction, based on remodeling of the upper forehead and the orbito-naso-frontal band (BONF). However, BONF reshaping is difficult to tailor to each individual child. In most cases, the surgeon performs the reshaping "freehand", without a template. The result is therefore subject to the surgeon's experience and judgment.

A surgical instrument (template) has been developed to guide the surgeon in the ideal reshaping of the BONF in patients with anterior craniostenosis (anterior plagiocephaly and trigonocephaly), according to each child's specific morphology.

The aim of EPBONF research is to evaluate the benefits of using this template on the symmetry and angle of the BONF.

ELIGIBILITY:
Inclusion Criteria:

* Children with anterior craniostenosis (organic trigonocephaly or anterior plagiocephaly), aged 4 to 24 months
* Procedure performed at Besançon University Hospital
* Written consent from both parents, or from one parent if there is only one, indicating that they have understood the purpose and procedures of the study, and that they agree to their child's participation in the study and to the study's requirements and restrictions.
* Affiliation with a French social security scheme or beneficiary of such a scheme.
* Pre-operative computed tomography scan and cone beam to measure the fronto zygomatic distance and naso-frontal angle in trigonocephaly, and to calculate the frontal process of the zygoma symmetry defect in organic anterior plagiocephaly.

Exclusion Criteria:

* Legal incapacity or limited legal capacity of parent(s)
* Subject is in the exclusion period of another study or is on the "national volunteer list".

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the performance of the medical device, for orbito-naso-frontal bandeau surgery, in the treatment of craniostenosis: evaluation of efficacy on orbito-naso-frontal bandeau conformation, angle and symmetry criteria. | 6 months after intervention
  Measurement of the frontal angle from scanned images and/or observation of symmetry or lack of symmetry of the orbito-naso-frontal bandeau :
  - frontal angle
Evaluating the performance of the medical device, for orbito-naso-frontal bandeau surgery, in the treatment of craniostenosis: evaluation of efficacy on orbito-naso-frontal bandeau conformation, angle and symmetry criteria. | 6 months after intervention
  Measurement of the frontal angle from scanned images and/or observation of symmetry or lack of symmetry of the orbito-naso-frontal bandeau :
  * symmetry for trigonocephaly
Evaluating the performance of the medical device, for orbito-naso-frontal bandeau surgery, in the treatment of craniostenosis: evaluation of efficacy on orbito-naso-frontal bandeau conformation, angle and symmetry criteria. | 6 months after intervention
  Measurement of the frontal angle from scanned images and/or observation of symmetry or lack of symmetry of the orbito-naso-frontal bandeau :
  - symmetry for plagiocephaly

IPD SHARING:
Plan to Share IPD: No